CLINICAL TRIAL: NCT03871413
Title: Can Benign Paroxysmal Positional Vertigo (BPPV) be Treated Faster and More Efficiently by Using a Mechanical Rotational Chair Compared to the Traditional Manual Repositioning Maneuvers?
Brief Title: TRV-chair vs Manual Repositioning Maneuver in Treatment of Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Dan Dupont Hougaard, MD, Associate Professor, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRV002
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: BPPV
Keywords: Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vestibular Diseases; Epley Maneuver; TRV-chair; Repositioning chair
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual repositioning maneuver (Active Comparator): Diagnostics and treatment of BPPV with manual repositioning maneuvers. In case of posterior canal involvement, Epley's maneuver will be used. In case of horizontal canal involvement, the log roll maneuver will be used.
  Interventions: Procedure: Manual repositioning maneuver
- Treatment in mechanical rotational chair (TRV-chair) (Experimental): Diagnostics and treatment of BPPV with the use of a TRV chair. In case of posterior canal involvement, Epley's maneuver will be used with the addition of 10 kinetic impulses in each position.
  In case of horizontal canal involvement, the log roll maneuver will be used with the addition of 10 kinetic impulses in each position.
  Interventions: Device: TRV-chair

INTERVENTIONS:
Device: TRV-chair — Repositioning maneuvers in TRV-chair
  Arms: Treatment in mechanical rotational chair (TRV-chair)
Procedure: Manual repositioning maneuver — Treatment with manual repositioning maneuver
  Arms: Manual repositioning maneuver

SUMMARY:
Comparison of treatment efficacy of a mechanical rotational chair (TRV-chair) vs. manual repositioning maneuvers in BPPV

DETAILED DESCRIPTION:
Open-label, randomized controlled trial comparing manual repositioning maneuvers with a mechanical rotational chair (TRV-chair) in diagnosing and treating BPPV. Patients with suspected BPPV will be randomized to either manual repositioning maneuvers or the TRV-chair.

ELIGIBILITY:
Inclusion Criteria:

* Characteristic (for BPPV) positional nystagmus
* Positive Dix-Hallpike
* Positive supine roll test
* Medical history compatible with BPPV

Exclusion Criteria:

* Treatment in TRV-chair within the last 6 months
* Exclusion of BPPV diagnosis
* Lack of treatment cooperation
* Known cerebral aneurism or cerebral hemorrhage
* Diagnosed and treated for BPPV within the past month
* Treatment with sedating anti-histamines within the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Number of treatments | 2 years
  Number of treatment necessary to achieve resolution of vertigo and nystagmus
Treatment success after first treatment | 2 years
  Number of subjects achieving resolution of vertigo and nystagmus after one treatment

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI) questionnaire | 2 years
  Comparison of pre-treatment score and post-treatment score
Adverse events | 2 years
  Registration of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dan D Hougaard, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Otolaryngology, Head & Neck Surgery and Audiology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No